CLINICAL TRIAL: NCT02035579
Title: Aerobic Training for Management of Post-Concussion Syndrome in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPR112665
Record Dates: First submitted 2013-09-05; First posted 2014-01-14 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Concussion; Post-concussion Syndrome; Sports Injury
Keywords: concussion; mild traumatic brain injury; post-concussion syndrome; adolescents; sports injury; aerobic training; stretching training
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Athletic Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Training Intervention (Experimental): Children with PCS who are eligible for the study will be randomized to a progressive, sub-symptom exacerbation, cycling aerobic training intervention or stretching comparison intervention. Children with PCS that meet criteria for the intervention trial will complete a baseline evaluation followed by a one week run-in-period (week 0-1) prior to their first intervention visit. After the initial intervention visit, weekly visits will be completed for at least 6 additional weeks (i.e., at least 6 weeks of aerobic training). An individualized home exercise program 5-6 days per week will also be developed. Children will be provided with a home stationary cycle to complete the home program.
  Interventions: Behavioral: Aerobic Training Intervention
- Stretching Intervention (Experimental): Children in the stretching intervention will complete a series of full body stretches of the shoulders, arms, chest, back, legs, and feet 5-6 days per week and will return weekly to review the stretching program. The minimum duration of the stretching intervention will also be 6 weeks
  Interventions: Behavioral: Stretching Intervention

INTERVENTIONS:
Behavioral: Aerobic Training Intervention
  Arms: Aerobic Training Intervention
Behavioral: Stretching Intervention
  Arms: Stretching Intervention

SUMMARY:
Sports-related concussions are common in adolescent-athletes. Prolonged recovery after concussion or post-concussion syndrome (PCS) is a public health problem. This project will determine the effectiveness of an aerobic exercise program for management of PCS and it will evaluate the influence of exercise on biologic correlates of PCS.

DETAILED DESCRIPTION:
Concussion or mild traumatic brain injury (mTBI) is a public health problem and it is imperative that efficacious treatment protocols be developed to reduce the morbidity associated with PCS in adolescents. In adolescent athletes, timely return of normal neurocognitive function and return to sports safely is critical to normal development. The proposed study will fill a critical gap by systematically evaluating the potential efficacy of an aerobic training intervention for management of PCS in adolescents. To our knowledge, this will be the first randomized controlled study to evaluate the efficacy of aerobic training for treatment of PCS in adolescents as soon as four weeks after injury. The study will also improve our understanding of the pathophysiology of PCS and the biologic influence of aerobic training on PCS. The proposed study will fill a critical gap and inform the development of larger studies to assess the efficacy, and if proven efficacious, optimize the timing and intensity of aerobic training treatment protocols, thus transforming the care and limiting the adverse public impact of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 12 to 17 years
* Experienced a concussion 4 to 16 weeks prior to enrollment
* Experiencing persistent post-concussion symptoms

Exclusion Criteria:

* Sustained a moderate to severe head injury, head injury more severe than concussion or required an overnight hospital stay
* Younger than 12 years of age when beginning the study.
* Older than 17 years of age when beginning the study.
* Do not live with a parent/guardian.
* Injured more than 16 weeks ago.
* Do not speak or read English.
* Diagnosed with a developmental disability.
* Neurological impairment, cognitive disorders, genetic disorders, metabolic disorders, blood disorder, cardiovascular problem/disease, and/or cancer.
* Inpatient admission for a psychiatric disorder within the past 12 months.
* Taking beta-blockers, anti-depressants, and/or anti-epileptic medications that cannot be discontinued while participating in the study.
* Cardiovascular condition that would preclude participation in the training protocol.
* Any condition that precludes magnetic resonance imaging (MRI).
* Females that are pregnant or become pregnant during the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in post-concussive symptoms at 10 week follow up | 1 year

SECONDARY OUTCOMES:
Change from baseline in cognitive functioning at 10 week follow up | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Brad Kurowski, MD, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Gladstone E, Narad ME, Hussain F, Quatman-Yates CC, Hugentobler J, Wade SL, Gubanich PJ, Kurowski BG. Neurocognitive and Quality of Life Improvements Associated With Aerobic Training for Individuals With Persistent Symptoms After Mild Traumatic Brain Injury: Secondary Outcome Analysis of a Pilot Randomized Clinical Trial. Front Neurol. 2019 Sep 18;10:1002. doi: 10.3389/fneur.2019.01002. eCollection 2019. PMID 31620073
- [Derived] Kurowski BG, Hugentobler J, Quatman-Yates C, Taylor J, Gubanich PJ, Altaye M, Wade SL. Aerobic Exercise for Adolescents With Prolonged Symptoms After Mild Traumatic Brain Injury: An Exploratory Randomized Clinical Trial. J Head Trauma Rehabil. 2017 Mar/Apr;32(2):79-89. doi: 10.1097/HTR.0000000000000238. PMID 27120294